CLINICAL TRIAL: NCT02767193
Title: Safety and Immunogenicity of a Vaccine Dendritic Cell-based Pulsed With Autologous Heat-inactivated HIV in HIV-1 Infected Patients. Prospective, Randomized, Partially Blinded Study
Brief Title: Safety and Immunogenicity of a Vaccine Dendritic Cell-based Pulsed With Autologous Heat-inactivated in HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCV3/RisVac04; 2015-001795-22 (EudraCT Number)
Record Dates: First submitted 2016-04-22; First posted 2016-05-10 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- DCV3 (Experimental): Autologus differentiated adult dendritic cells from monocytes of peripheral blood non expanded pulsed with autologous inactivated HIV virus
  Interventions: Biological: DCV3
- DCV3 with PEG-INF (Experimental): Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded pulsed with autologous inactivated HIV virus with PEG-INF
  Interventions: Biological: DCV3 with PEG-INF
- CD placebo (Placebo Comparator): Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded
  Interventions: Biological: Placebo
- CD placebo + PEG-INF (Placebo Comparator): Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded with PEG-INF
  Interventions: Biological: Placebo with PEG-INF

INTERVENTIONS:
Biological: DCV3 — Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded pulsed with autologous inactivated HIV virus.
  Patients will receive three immunizations of dendritic cells during weeks 0, 2 and 4
  Arms: DCV3
Biological: DCV3 with PEG-INF — Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded pulsed with autologous inactivated HIV virus with PEG_INF Patients will receive three immunizations of dendritic cells during weeks 0, 2 and 4 and INF during weeks 4,5 and 6
  Arms: DCV3 with PEG-INF
Biological: Placebo — Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded Patients will receive three immunizations saline + 1% albumin during weeks 0, 2 and 4
  Arms: CD placebo
Biological: Placebo with PEG-INF — Autologous differentiated adult dendritic cells from monocytes of peripheral blood non expanded with PEG_INF Patients will receive three immunizations saline + 1% albumin during weeks 0, 2 and 4 and INF during weeks 4,5 and 6.
  Arms: CD placebo + PEG-INF

SUMMARY:
single-center, national clinical trial, phase I, randomized (1: 1: 1: 1), prospective, placebo-controlled, partially masked, parallel group. Patients will be assigned to one of the following four arms: 3 immunizations of dendritic cells / 3 immunizations of dendritic cells with pegylated interferon + / 3 immunizations of placebo / 3 immunizations of placebo with pegylated interferon.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years of age;
2. Voluntarily sign informed consent;
3. Men or women with a negative pregnancy test before inclusion in the study;
4. HIV infection tested (with positive antibodies to HIV-1 and a detectable viral load);
5. Patient must be on stable treatment with cART at least 1 year
6. The average of all measurements of CD4 during the year before starting cART should be equal or greater than 350 cells / mm3
7. The number of CD4 + at enrollment must be equal or greater than 450 cells / mm3;
8. Plasma HIV viral load undetectable at least 6 months before the inclusion in the study, at least two determinations (occasional blips above the undetectable level are allowed).

Exclusion Criteria:

1. Treatment with suboptimal regimen (less than 3 antiretroviral drugs) before starting cART;
2. History of C CDC events;
3. Interruption of cART during the inclusion in the study;
4. Pregnancy woman or becoming pregnant in the next months;
5. Active opportunistic infections, or any active infection or cancer within 30 days prior to the screening visit;
6. Therapy with immunomodulatory agents, including cytokines (eg IL-2) and gamma globulins or chemotherapy within 90 days prior to the screening visit;
7. Use of anticoagulant medication;
8. Use of any investigational drug within 90 days prior to study entry;
9. Virological failure prior to antiretroviral treatment and / or mutations that confer resistance to antiretroviral drugs;
10. Uncontrolled psychiatric disorder;
11. Platelet count <80,000 / mm3;
12. Values ??of hemoglobin <12g / dL;
13. Patients with active uncontrolled autoimmune diseases;
14. Using contraindicated drugs in accordance with the Summary of Product Specifications of pegylated interferon;
15. Childbearing, or potential childbearing not using highly effective contraception;
16. Any other problem that according to the investigator could interfere with the evaluation of the objectives.
17. Any contraindication for the use of interferon peg in accordance with the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05; Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Number of Participants with adverse events of grade 3 or higher | 28 weeks
  * Local adverse events of grade 3 or higher (pain and skin reactions including induration)
  * Systemic adverse events of grade 3 or higher (fever, chills, headache, nausea, vomiting, malaise and myalgia)
  * Clinical or laboratory confirmed grade 3 or higher on physical examination or retests adverse events Any event attributable to the vaccine involving a discontinuation of vaccination regime.
Virological | 12 weeks
  Proportion of patients with undetectable viral load (<37 copies / mL) at 12 weeks

SECONDARY OUTCOMES:
Number of adverse events grade 1 and 2 within 14 days after each immunization (weeks 2, 4 and 6) | 6 weeks
Changes in the specific immune response | 28 weeks
  Measured by ELISPOT visits in weeks 2, 4, 8, 12, 16 and 28 compared to baseline and screening for dendritic cell vaccine and pegylated interferon.
Changes in levels of viral reservoir. | 28 weeks
  Measure the proviral DNA visits in the weeks -44, -36, 4, 8, 12, 16 and 28 compared to baseline and screening.
Proportion of patients with changes in any value of the levels of inflammatory markers, microbial translocation and immune activation | 28 weeks
  In visits at weeks 4, 16 and 28 compared compared to baseline and screening
Proportion of patients with viral rebound | 15 days
  Two consecutive obtaining measurements of plasma viral load> 37 copies / mL separated by at least 15 days after discontinuation of antiretroviral therapy.
Proportion of patients with autoimmunity markers induced by the vaccine as measured by: antithyroid antibodies (antithyroglobulin, antithyroid peroxidase), antinuclear antibodies, antiphospholipid antibodies and rheumatoid factors. | 16 weeks
  Evaluation on autoimmunity with antithyroid antibodies (antithyroglobulin, antithyroid peroxidase), antinuclear antibodies, antiphospholipid antibodies and rheumatoid factor at screening, baseline and week 16.
Changes in the transcriptome of patients visits weeks 4, 16 and 28 compared to baseline (week -12) | 28 weeks
  Weeks 4, 16 and 28 compared to baseline
Evaluation of the specific immune response trought IFN-gamma production in vitro at screening and baseline | week 0
  Proportion of patients with IFN-gamma production in vitro measured by ELISPOT at screening and baseline
Evaluation of the specific immune response thought dendritic cell maturation markers in vitro at screening and baseline | week 0
  Proportion of patients with dendritic cell maturation markers in vitro measured by flow cytometry at screening and baseline
Evaluation of the specific immune response thought T-cell proliferation in vitro at screening and baseline | week 0
  Proportion of patients with T-cell proliferation in vitro measured by CFSE (carboxyfluorescein succinimidyl ester) at screening and baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic, Barcelona, España, Spain

REFERENCES:
- [Derived] Leal L, Couto E, Sanchez-Palomino S, Climent N, Fernandez I, Miralles L, Romero Y, Gonzalez T, Maleno MJ, Pano B, Pich J, Nicolau C, Gatell JM, Plana M, Garcia F; DCV3-RISVAC04 Study Group. Effect of Intranodally Administered Dendritic Cell-Based HIV Vaccine in Combination With Pegylated Interferon alpha-2a on Viral Control Following ART Discontinuation: A Phase 2A Randomized Clinical Trial. Front Immunol. 2021 Nov 11;12:767370. doi: 10.3389/fimmu.2021.767370. eCollection 2021. PMID 34858423